CLINICAL TRIAL: NCT07270562
Title: ORbital Atherectomy for Lesion Preparation in Patients With Chronic Limb-threatening ischEmia
Acronym: ORACLE
Status: Not yet recruiting | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: ORACLE
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Limb Threatening Ischemia; Chronic Limb-Threatening Ischemia
Keywords: CLTI; Peripheral artery disease; Orbital atherectomy; Observational cohort study; Chronic limb ischemia; Critical limb-threatening ischemia; Calcified peripheral artery lesions; Vessel preparation; Femoropopliteal arteries; Infrapopliteal arteries; OA; Atherectomy for calcified lesions
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult CLTI patients with femoropopliteal or infrapopliteal calcified lesions: Eligible patients are those who will undergo OA prior to any adjunctive endovascular procedure
  Interventions: Device: Stealth 360™ Peripheral Orbital Atherectomy System from Abbott

INTERVENTIONS:
Device: Stealth 360™ Peripheral Orbital Atherectomy System from Abbott — The Stealth 360™ Peripheral Orbital Atherectomy System uses a diamond-coated, eccentrically mounted crown with bi-directional capabilities that treat a wide range of vessels, enabling single device treatment of multiple lesions and vessel sizes.
  Other Names: Orbital Atherectomy; Orbital Atherectomy System

SUMMARY:
ORACLE is a Europe-wide study that will follow 250 people with critical limb-threatening ischemia (CLTI). It aims to see how well orbital atherectomy (OA) works in real-life practice. OA is a procedure that uses a tiny spinning tool to gently remove hard calcium from inside an artery, helping to open the vessel so other treatments-like balloons or stents-can work better. The study focuses on people who have heavily calcified arteries in the femoropopliteal or infrapopliteal areas of the leg.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford classification category ≥4;
2. Treatment of femoropopliteal or infrapopliteal calcified lesions with OA using the Stealth 360 peripheral OA System;
3. Calcification of target lesions must be visible on fluoroscopy or CT-angiography;
4. Patients competent and willing to provide informed consent.

Exclusion Criteria:

1. Minors and other vulnerable populations who may not be able to give informed consent freely or for whom participation is not essential to the study (incapacitated and unconscious individuals, persons deprived of liberty, pregnant and breastfeeding women, etc.);
2. Inadequate inflow (>30% stenosis) following optimization;
3. Insufficient direct outflow (less than 1 run-off vessel);
4. Endovascular procedure(s) on the treatment site within 4 weeks before index procedure;
5. Patients planned to receive an above ankle amputation of the target limb;
6. Patients enrolled in RESCUE (ClinicalTrials.gov ID NCT07270575).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CLTI patients with femoropopliteal or infrapopliteal calcified lesions treated with OA using the Stealth 360 Peripheral OA System for vessel preparation prior to any adjunctive endovascular procedure.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Number of lesions with ≤30% residual stenosis after completion of full planned procedure | Immediately after procedure completion
  Defined as residual stenosis ≤30%, immediately after completion of full planned procedure (OA + any planned adjunctive intervention(s)).

SECONDARY OUTCOMES:
Number of lesions with ≤30% residual stenosis after any unplanned endovascular intervention(s) | Immediately after procedure completion
  Defined as residual stenosis ≤30% immediately after completion of additional unplanned endovascular intervention(s) (any endovascular procedure that was not part of the primary procedure plan).
Need for unplanned bailout stenting | Immediately after procedure completion
  Defined as any stent placement that was not part of the primary procedure plan.
Number of participants free from Clinically-Driven Target Lesion Revascularization (CD-TLR) | 12 and 24 months
  Defined as freedom from any endovascular re-intervention to the target lesion (± 10 mm) or surgical bypass performed because of restenosis or occlusion of the target lesion.
CD-TLR-free survival | Until the end of the follow-up period of 2 years
  Defined as time between first OA procedure and any endovascular re-intervention to the target lesion (± 10 mm) or surgical bypass performed because of restenosis or occlusion of the target lesion.
Clinical response using Rutherford classification categories | 12 and 24 months
  The Rutherford classification is a clinical scale used to categorize the severity of peripheral arterial disease: Category 0 = asymptomatic; Category 1 = mild claudication; Category 2 = moderate claudication; Category 3 = severe claudication; Category 4 = ischemic rest pain; Category 5 = minor tissue loss; Category 6 = severe tissue loss.
Wound status | 12 and 24 months
  Defined as healing status of the dominant ischemic wound of the target limb (complete, partial, unchanged, worsening).
Freedom from amputation of the target limb | 12 and 24 months
  Defined as absence of any amputation of the target limb (above ankle).
Amputation-free survival | Until the end of the follow-up period of 2 years
  Defined as time between first OA procedure and above-ankle amputation of the target limb.
Overall survival | Until the end of the follow-up period of 2 years
  Defined as the time between the first OA procedure and death of any cause.
Patient-reported health-related quality-of-life | Baseline, 6, 12 and 24 months post treatment
  Measured by Vascular Quality of Life Questionnaire - 6 items (VascuQol-6), which is a short patient-reported outcome measure (PROM), used to assess health-related quality of life in people with PAD. It consists of 6 questions, each scored from 1 to 7, with 1 as the worst possible quality of life and 7 as the best possible quality of life. Higher overall scores reflect better quality of life for patients with PAD.
Frequency and severity of procedural complications and other adverse events | Within 30 days after the OA procedure
  Grading according to the classification system of the Cardiovascular and Interventional Radiological Society of Europe.
Clinical response using ankle-brachial index (ABI) | 12 and 24 months
  The ankle-brachial index (ABI) is a non-invasive measure calculated as the ratio of systolic blood pressure at the ankle to systolic blood pressure at the arm. ABI categories commonly used to classify peripheral arterial disease are: >1.40 = non-compressible arteries; 1.00-1.40 = normal; 0.91-0.99 = borderline; 0.41-0.90 = mild to moderate peripheral arterial disease; <0.40 = severe peripheral arterial disease.
Clinical response using toe pressure | 12 and 24 months
  The toe pressure test measures distal limb perfusion by recording systolic pressure at the toe. In CLTI patients, toe pressure ≤30 mmHg is commonly used to indicate severe ischemia, while values >30 mmHg suggest better perfusion.
Clinical response using WIfi (wound, ischemia and foot infection) score | 12 and 24 months
  The WIfI classification is a staging system used to assess CLTI based on wound extent, ischemia severity, and foot infection. Each component is graded from 0 (none) to 3 (severe). Lower WIfI scores indicate a lower risk of limb loss and a lesser urgency for revascularization, whereas higher scores indicate greater disease severity, higher amputation risk, and greater potential benefit from revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Grözinger, Prof. Dr. med., Study Chair — SLK Kliniken Heilbronn GmbH; Marianne Brodmann, Univ.-Prof. Dr. med., Study Chair — Medizinische Universität Graz; Raghu Lakshminarayan, Dr, Study Chair — Hull University Teaching Hospitals NHS Trust; Stefan Müller-Hülsbeck, Prof. Dr. med., Study Chair — DIAKO Krankenhaus gGmBH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nordanstig J, Wann-Hansson C, Karlsson J, Lundstrom M, Pettersson M, Morgan MB. Vascular Quality of Life Questionnaire-6 facilitates health-related quality of life assessment in peripheral arterial disease. J Vasc Surg. 2014 Mar;59(3):700-7. doi: 10.1016/j.jvs.2013.08.099. Epub 2013 Dec 15. PMID 24342060
- [Background] Filippiadis DK, Binkert C, Pellerin O, Hoffmann RT, Krajina A, Pereira PL. Cirse Quality Assurance Document and Standards for Classification of Complications: The Cirse Classification System. Cardiovasc Intervent Radiol. 2017 Aug;40(8):1141-1146. doi: 10.1007/s00270-017-1703-4. Epub 2017 Jun 5. PMID 28584945